CLINICAL TRIAL: NCT03212833
Title: Impact of Insulin Resistance on Therapeutic Response for Oral Treatment of Chronic Hepatitis C Virus Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hosny Sayed, dr, Assiut University
Other Study IDs: 17200093
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: fasting serum insulin — fasting serum insulin in chronic hepatitis C patients

SUMMARY:
Globally, approximately 170 million people are infected with hepatitis C virus (HCV); 350,000 deaths each year are caused by HCV infection (Perz,et al, 2006).The Egyptian Demographic Health Survey (EDHS), across sectional survey including hepatitis C virus (HCV)biomarkers, was conducted in 2008 on a large nationally representative sample (El-Zanaty F, et al 2009). It estimated HCV prevalence among the 15-59 years age group to be 14.7% (El-Zanaty F, et al 2009).Accordingly, Egypt has the highest HCV prevalence in the world (Lavanchy D, 2011), ( Shepard CW,et al 2005)..Interferon (INF)-free regimens of combined directly acting antivirals (DAAs) have shown improved efficacy and tolerability compared with interferon (IFN)-containing regimens, and they have become the standard of care for treatment of HCV genotype-1 (HCV-1)(Afdhal, et al, 2014).Insulin resistance is a state in which a given concentration of insulin produces a less-than-expected biological effect. The prevalence of type 2 diabetes mellitus in hepatitis C in cirrhotic patients is 27.3% which is higher than among non-cirrhotic hepatitis C patients (17.5%)(Romero-Gómez, 2006). HCV promotes insulin resistance and insulin resistance induces interferon resistance, steatosis and fibrosis progression in a genotype-dependent manner.In HCV-1, insulin resistance decreases sustained response rate, and increase the risk for the development of steatosis and fibrosis progression, However, the impact of insulin resistance in other genotypes seems not achieve enough importance to impair sustained response, probably due to the high sensitivity to peginterferon. The treatment of insulin resistance, decreasing hyperinsulinemia, could improve sustained response rate in patients with chronic HCV-1 infection when treated with peginterferon plus ribavirin(Romero-Gómez,2006).

Objectives: we aim to determine the prevalence of insulin resistance among the patients with chronic hepatitis C virus( HCV) infection and to explore the association between insulin resistance and therapeutic response by comparing the insulin resistance among responders and non-responders to oral treatment of chronic hepatitis C virus infection Patients and methods: The study is intended to include patients of chronic hepatitis C virus infection receiving oral treatment for one year period. All patients will have clinical evaluation, ultrasonographic examination, and laboratory investigations which include complete blood count, liver function tests, estimation of fasting serum glucose, fasting serum insulin, and determination of insulin resistance index.The patients will be selected according the selection criteria determined by the National Committee for Control of Viral Hepatitis (NCCVH).

ELIGIBILITY:
Inclusion Criteria:

* The study is intended to include patients with chronic HCV infection.

Exclusion Criteria:

* Presence of large risky esophageal varices (except after successful prophylactic banding).
* Uncontrolled ascites.
* Patients with hepatocellular carcinoma except after successful curative intervention (3 months after resection or successful loco-regional therapy).
* Child score of 8 or less.
* Total serum bilirubin of 5 mg/dL or less.
* Platelet count of 30000/mm3 or more.
* Hemoglobin level of 10 g/DL or more.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with chronic HCV infection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
fasting serum insulin | 10 minutes
  which is estimated fasting serum insulin in micro international unit per millileter

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt